CLINICAL TRIAL: NCT01738555
Title: An Open-label, 36-week Extension Study on Amdoxovir at 500 mg Bid or 300 mg Bid in Combination With Zidovudine and Lopinavir/Ritonavir in HIV-1 Treatment-experienced Subjects With M184I/V Mutation in Addition to 0-2 Confirmed Thymidine Analog Mutations.
Brief Title: A Safety and Efficacy Study of Amdoxovir in HIV-1 Treatment-experienced Subjects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: RFS Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFSP-AMDX-2012
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Human Immunodeficiency Virus Infection
Keywords: amdoxovir; zidovudine; HIV; HAART; antiretroviral
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — amdoxovir; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- amdoxovir 300 mg bid (Experimental): in combination with zidovudine 300 mg bid and lopinavir/ritonavir (400 mg/100 mg bid) for 36 weeks.
  Interventions: Drug: amdoxovir 300 mg bid
- amdoxovir 500 mg bid (Experimental): in combination with zidovudine 300 mg bid and lopinavir/ritonavir (400 mg/100 mg bid) for 36 weeks.
  Interventions: Drug: amdoxovir 500 mg bid

INTERVENTIONS:
Drug: amdoxovir 300 mg bid — 2 x 150 mg capsules bid
  Other Names: DAPD; AMDX
  Arms: amdoxovir 300 mg bid
Drug: amdoxovir 500 mg bid — 2 x 250 mg capsules bid
  Other Names: DAPD; AMDX
  Arms: amdoxovir 500 mg bid

SUMMARY:
This study is an open-label extension of RFSP-AMDX-2010 study for those subjects who received treatment with amdoxovir (300 mg or 500 mg twice daily) for 12 weeks and benefited from it. This study will examine the safety and efficacy of the investigational HIV drug, amdoxovir (300 mg and 500 mg bid doses; N = up to 30) in combination with zidovudine and lopinavir/ritonavir for 36 weeks.

Subjects will continue to receive either amdoxovir 300 mg twice daily or amdoxovir 500 mg twice daily, each in combination with zidovudine 300 mg twice daily and lopinavir/ritonavir (400 mg/100 mg twice daily) for additional 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed Study RFSP-AMDX-2010 and received treatment with amdoxovir (500 mg bid or 300 mg bid) for 12 weeks before entry into study RFSP-AMDX-2012.
* Must have maintained ≥ 1.0 log10 copies/mL from baseline at Week 12 in Study RFSP-AMDX-2010.
* Must not have had any serious adverse experience since enrollment in Study RFSP-AMDX-2010, whether or not considered to be study drug-related.

Exclusion Criteria:

* Subjects who require ongoing therapy of nephrotoxic drugs or competitors of renal excretion.
* Subjects who require therapy with hematologic, bone marrow suppressive or cytotoxic agents.
* Subjects who require medications that are highly dependent on CYP3A for clearance and for which elevated plasma concentrations are associated with life-threatening adverse events.
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulations.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
HIV-1 viral load | up to 48 Weeks

SECONDARY OUTCOMES:
Incidence of adverse events | up to 48 Weeks
Changes in Immunologic Function (CD4 cell counts) | from baseline to Weeks 18, 24, 30, 36, 42, 48

CONTACTS AND LOCATIONS:
Overall Officials: Luz Pascual, MD MPH, Study Director — RFS Pharma, LLC